CLINICAL TRIAL: NCT03947788
Title: One Key Question-System Team Patient: A Pilot Study Phase II
Brief Title: One Key Question: Pilot Study at NorthShore
Acronym: OKQ2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Endeavor Health (Other)
Collaborators: University of Chicago (Other)
Responsible Party: Principal Investigator, Emily White VanGompel, Clinical Assistant Professor, Endeavor Health
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: EH18-343
Record Dates: First submitted 2019-05-09; First posted 2019-05-13 (Actual); Results first posted 2021-11-09 (Actual); Last update posted 2021-12-03 (Actual); Status verified 2021-12

CONDITIONS: Reproductive Health

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional Practices (Experimental): These clinics, including physicians, clinical and administrative staff, will receive the One Key Question training program, delivered by Power to Decide, via an in-person group training session.
  Interventions: Behavioral: OKQ Training Program
- Control Practices (No Intervention): These clinics will not receive the OKQ training program during the study period. They will have the opportunity to receive the training after the study period is over.

INTERVENTIONS:
Behavioral: OKQ Training Program — The OKQ training program helps clinicians more efficiently meet the needs of women's pregnancy intentions and provide evidence-based care.
  Arms: Interventional Practices

SUMMARY:
This study is a pilot assessment of whether practices that implement the One Key Question® (OKQ) pregnancy intention screening tool will demonstrate differences in patient-reported receipt of preconception and/or contraceptive counseling, compared to practices that provide usual care. In Phase I, the study team surveyed patients at six practices within NorthShore University HealthSystem to establish baseline rates of counseling. Phase II assesses the effects of the OKQ tool on patient care, and half of participating sites are randomly chosen as intervention sites and exposed to the OKQ tool. After the intervention practices implement OKQ, patients will be surveyed at both intervention and control (usual care) practices to measure changes in preconception and contraceptive care.

DETAILED DESCRIPTION:
Effectively delivered preconception counseling leads to healthier pregnancy behaviors. However, many clinicians miss opportunities to provide this counseling due to a lack of processes in place to provide this counseling and access to evidence based care once the need is identified. The purpose of this study is to build upon baseline data collected on pregnancy intention and receipt of contraceptive and preconception counseling. Half of the study practices will be randomly selected to receive comprehensive One Key Question® Training through the nonprofit Power To Decide. These practices have already displayed interest in taking part in this intervention.The training will act as our intervention, and will be given to help improve the quality of preconception and contraceptive counseling in Primary Care and Obstetrics/Gynecology. All of the participating practices will then be surveyed again to determine changes in contraception and preconception counseling. After patient data collection is complete, a research assistant will return to each practice to collect surveys from clinicians and staff (this includes: physicians, nurses, medical assistants, patient support associates, or anyone that participated in the OKQ training) at the intervention practices to assess the experience of implementing OKQ and their perceptions of its utility for patients. Following the Phase II collection of surveys, the remaining control practices will be given the option to receive Power To Decide training.

ELIGIBILITY:
Inclusion Criteria:

* Female
* 18-49 years old
* Receiving either primary or obstetric/gynecology care at one of the study clinics

Exclusion Criteria:

* Male
* Pregnant
* <18 years old >49 years old

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Female
Enrollment: 143 (Actual)
Dates: Start 2019-01-17 (Actual); Primary Completion 2021-01-06 (Actual); Study Completion 2021-01-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Emily White VanGompel, MD, MPH, Principal Investigator — Endeavor Health
Locations (1):
- Northshore University HealthSystem, Evanston, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Williams L, Zapata LB, D'Angelo DV, Harrison L, Morrow B. Associations between preconception counseling and maternal behaviors before and during pregnancy. Matern Child Health J. 2012 Dec;16(9):1854-61. doi: 10.1007/s10995-011-0932-4. PMID 22173331
- [Background] Dehlendorf C, Henderson JT, Vittinghoff E, Grumbach K, Levy K, Schmittdiel J, Lee J, Schillinger D, Steinauer J. Association of the quality of interpersonal care during family planning counseling with contraceptive use. Am J Obstet Gynecol. 2016 Jul;215(1):78.e1-9. doi: 10.1016/j.ajog.2016.01.173. Epub 2016 Jan 28. PMID 26827879
- [Background] Dehlendorf C, Krajewski C, Borrero S. Contraceptive counseling: best practices to ensure quality communication and enable effective contraceptive use. Clin Obstet Gynecol. 2014 Dec;57(4):659-73. doi: 10.1097/GRF.0000000000000059. PMID 25264697
- [Background] Shannon GD, Alberg C, Nacul L, Pashayan N. Preconception healthcare and congenital disorders: systematic review of the effectiveness of preconception care programs in the prevention of congenital disorders. Matern Child Health J. 2014 Aug;18(6):1354-79. doi: 10.1007/s10995-013-1370-2. PMID 24091886
- [Background] Temel S, van Voorst SF, Jack BW, Denktas S, Steegers EA. Evidence-based preconceptional lifestyle interventions. Epidemiol Rev. 2014;36:19-30. doi: 10.1093/epirev/mxt003. Epub 2013 Aug 28. PMID 23985430
- [Background] Mohllajee AP, Curtis KM, Morrow B, Marchbanks PA. Pregnancy intention and its relationship to birth and maternal outcomes. Obstet Gynecol. 2007 Mar;109(3):678-86. doi: 10.1097/01.AOG.0000255666.78427.c5. PMID 17329520
- [Background] Gavin L, Moskosky S, Carter M, Curtis K, Glass E, Godfrey E, Marcell A, Mautone-Smith N, Pazol K, Tepper N, Zapata L; Centers for Disease Control and Prevention (CDC). Providing quality family planning services: Recommendations of CDC and the U.S. Office of Population Affairs. MMWR Recomm Rep. 2014 Apr 25;63(RR-04):1-54. PMID 24759690
- [Background] Bello JK, Rao G, Stulberg DB. Trends in contraceptive and preconception care in United States ambulatory practices. Fam Med. 2015 Apr;47(4):264-71. PMID 25853596
- [Background] Bellanca HK, Hunter MS. ONE KEY QUESTION(R): Preventive reproductive health is part of high quality primary care. Contraception. 2013 Jul;88(1):3-6. doi: 10.1016/j.contraception.2013.05.003. Epub 2013 May 11. No abstract available. PMID 23773527
- [Background] Allen D, Hunter MS, Wood S, Beeson T. One Key Question(R): First Things First in Reproductive Health. Matern Child Health J. 2017 Mar;21(3):387-392. doi: 10.1007/s10995-017-2283-2. PMID 28220337
- [Background] Frayne DJ, Verbiest S, Chelmow D, Clarke H, Dunlop A, Hosmer J, Menard MK, Moos MK, Ramos D, Stuebe A, Zephyrin L. Health Care System Measures to Advance Preconception Wellness: Consensus Recommendations of the Clinical Workgroup of the National Preconception Health and Health Care Initiative. Obstet Gynecol. 2016 May;127(5):863-872. doi: 10.1097/AOG.0000000000001379. PMID 27054935
- [Background] Rocca CH, Ralph LJ, Wilson M, Gould H, Foster DG. Psychometric Evaluation of an Instrument to Measure Prospective Pregnancy Preferences: The Desire to Avoid Pregnancy Scale. Med Care. 2019 Feb;57(2):152-158. doi: 10.1097/MLR.0000000000001048. PMID 30550399
- [Derived] Ferketa M, Schueler K, Song B, Carlock F, Stulberg DB, White VanGompel E. Facilitators of and Barriers to Successful Implementation of the One Key Question(R) Pregnancy Intention Screening Tool. Womens Health Rep (New Rochelle). 2022 Mar 8;3(1):326-334. doi: 10.1089/whr.2021.0100. eCollection 2022. PMID 35415707

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Interventional Practices | Control Practices
Started | 69 | 74
Completed | 69 | 74
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Baseline data was based upon the characteristics of 4 clinics. The 4 clinics continued their participation for the duration of Phase 2 of the study. The interventional as well as the control group each consisted of one family medicine practice, and one OB/GYN practice. At baseline, a total of 69 subjects participated in the interventional group, and a total of 74 subjects participated in the control group.
Groups:
- Interventional Practices: The staff at these two clinics which included physicians, clinical and administrative staff; received the One Key Question in-person training program, delivered by Power to Decide.
  OKQ Training Program: The OKQ training program helps clinicians more efficiently meet the needs of women's pregnancy intentions and provide evidence-based care.
- Control Practices: These two clinics did not receive the One Key Question training program during the study period. They were offered the training after the study period was over.
- Total: Total of all reporting groups
Arm/Group | Interventional Practices | Control Practices | Total
Number analyzed (Participants) | 69 | 74 | 143
Age, Customized [Count of Participants; unit: Participants]
  Count of participants | 69 | 74 | 143
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 69 | 74 | 143
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 14 | 11 | 25
  Not Hispanic or Latino | 46 | 58 | 104
  Unknown or Not Reported | 9 | 5 | 14

OUTCOME MEASURES:

1. Primary Outcome: Receipt of Any Reproductive Health Counseling
Description: Among patients with potential to become pregnant, percent of respondents who received any reproductive health counseling. Counts as "Yes" for this outcome if they received any contraceptive counseling or any preconception counseling.
Time Frame: After the clinic has implemented OKQ for at least 4 weeks
Population: The population analyzed included patients with the ability to get pregnant that were between the ages of 18-49 years old. Patients that reported experiencing menopause, hysterectomy, or sterilization were excluded from analysis. Patients that were pregnant were not eligible for participation.
Measure: Count of Participants; unit: Participants
Groups:
- Interventional Practices: Patient recruitment for the intervention group occurred at the two clinics (one Family Medicine, one OB/GYN), that participated in the intervention (received the One Key Question training program).
  Patients at the intervention practices were surveyed to determine if there was an improved rate of received contraception counseling, following each clinic's implementation of the intervention for 4-6 weeks.
- Control Practices: Patient recruitment for the control group occurred at the two clinics (one Family Medicine, one OB/GYN), that did not participate in the intervention (did not receive One Key Question training program).
  Patients at the control practices were surveyed to demonstrate that contraception counseling rates remained unchanged at clinics not receiving the One Key Question training program.
Arm/Group | Interventional Practices | Control Practices
Number analyzed (Participants) | 69 | 74
Participants | 54 | 38

2. Secondary Outcome: Receipt of Contraceptive Counseling
Description: Among patients with potential to become pregnant, the rate of survey respondents who received any contraceptive counseling.
Time Frame: After the clinic has implemented OKQ for at least 4 weeks
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Groups:
- Interventional Practices: Patient recruitment for the intervention group occurred at the two clinics (one Family Medicine, one OB/GYN), that participated in the intervention (did not receive One Key Question training program).
  Patients at the intervention practices were surveyed to determine if there was an improved rate of received contraception counseling, following each clinic's implementation of the intervention for 4-6 weeks.
Arm/Group | Interventional Practices | Control Practices
Number analyzed (Participants) | 69 | 74
Participants | 45 | 33

3. Secondary Outcome: Receipt of Preconception Counseling
Description: Among patients with potential to become pregnant, percent of respondents who received any preconception counseling.
Time Frame: After the clinic has implemented OKQ for at least 4 weeks
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Groups:
- Interventional Practices, Clinics Receiving One Key Question Training: Patient recruitment for the intervention group occurred at the two clinics (one Family Medicine, one OB/GYN), that participated in the intervention (received One Key Question training program).
  Patients at the intervention practices were surveyed to determine if there was an improved rate of received preconception counseling, following each clinic's implementation of the intervention for 4-6 weeks.
- Control Practices, Clinics Not Receiving One Key Question Training: Patient recruitment for the control group occurred at the two clinics (one Family Medicine, one OB/GYN), that did not participate in the intervention (did not receive One Key Question training program).
  Patients at the control practices were surveyed to demonstrate that preconception counseling rates remained unchanged at clinics not receiving the One Key Question training program.
Arm/Group | Interventional Practices, Clinics Receiving One Key Question Training | Control Practices, Clinics Not Receiving One Key Question Training
Number analyzed (Participants) | 69 | 74
Participants | 26 | 13

4. Other Pre Specified Outcome: Patient Satisfaction With Overall Care
Description: This outcome measure can be described as the distribution of patient responses (extremely satisfied, very satisfied, satisfied, very dissatisfied, extremely dissatisfied) when asked about satisfaction with overall medical care during their visit. This outcome was measured as a count of patients that reported being very or extremely satisfied with the overall care provided at their visit that day.
Time Frame: After the clinic has implemented OKQ for at least 4 weeks.
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Groups:
- Interventional Practices: The intervention group consisted of two clinics (one Family Medicine, one OB/GYN), where physicians and staff received the One Key Question training program, delivered by Power to Decide, via an in-person group training session.
  OKQ Training Program: The OKQ training program helps clinicians more efficiently meet the needs of women's pregnancy intentions and provide evidence-based care.
  Patients at the two clinics were surveyed to determine if patient satisfaction increased following the clinics' implementation of the One Key Question program for 4-6 weeks.
- Control Practices: The control group consisted of two clinics (one Family Medicine, one OB/GYN), that did not receive the intervention (the One Key Question training program).
  Patients at the two clinics in the control group were surveyed to demonstrate that patient satisfaction remained unchanged among clinics not receiving the One Key Question training intervention.
Arm/Group | Interventional Practices | Control Practices
Number analyzed (Participants) | 69 | 74
Participants | 67 | 57

5. Other Pre Specified Outcome: Patient Satisfaction-Improving Their Health
Description: This outcome measure can be described as the distribution of patient responses (extremely satisfied, very satisfied, satisfied, very dissatisfied, extremely dissatisfied) when asked about satisfaction with the way their provider talked with them about improving their health.
  This outcome was measured as a count of patients that reported being very or extremely satisfied with the way their provider talked with them about improving their health.
Time Frame: After the clinic has implemented OKQ for at least 4 weeks
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Interventional Practices | Control Practices
Number analyzed (Participants) | 69 | 74
Participants | 64 | 54

ADVERSE EVENTS:
Description: All-cause Mortality, Serious, and Other [non-serious] Adverse Events were not monitored/assessed. This study was determined to be minimal risk with the potential for loss of confidentiality being the only risk to subjects. Monitoring subjects for All-cause Mortality, Serious, and Other Adverse Events was not required for this study.
Arm/Group | Interventional Practices | Control Practices
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2019-09-19): https://cdn.clinicaltrials.gov/large-docs/88/NCT03947788/Prot_003.pdf
  • Statistical Analysis Plan (2020-11-17): https://cdn.clinicaltrials.gov/large-docs/88/NCT03947788/SAP_004.pdf
  • Informed Consent Form (2018-01-23): https://cdn.clinicaltrials.gov/large-docs/88/NCT03947788/ICF_002.pdf